CLINICAL TRIAL: NCT03055481
Title: A Prospective Multicenter Non-inferiority Randomized Controlled Trial of the Irradiance Level of Phototherapy for Neonatal Jaundice
Brief Title: A Trial of the Irradiance Level of Phototherapy for Neonatal Jaundice
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: it was estimated that the recruitment of the planned number of patients could not be completed within further 5 years.
Sponsor: Nagoya University (Other)
Responsible Party: Principal Investigator, Yoshiaki Sato, Associate professor, Nagoya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-04-8
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Neonatal Jaundice
Keywords: neonatal jaundice; phototherapy; neonate
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High level irradiation (Active Comparator): High level irradiation: the target irradiance level is 30-35uW per square centimeter per nano-meter of wavelength.
  Interventions: Other: High irradiance level of phototherapy
- Low level irradiation (Experimental): Low level irradiation: the target irradiance level is 12-15uW per square centimeter per nano-meter of wavelength.
  Interventions: Other: Low irradiance level of phototherapy

INTERVENTIONS:
Other: High irradiance level of phototherapy — High irradiance level of phototherapy: the target irradiance level is 30-35uW per square centimeter per nanometer of wavelength.
  Arms: High level irradiation
Other: Low irradiance level of phototherapy — Low irradiance level of phototherapy: the target irradiance level is 12-15uW per square centimeter per nanometer of wavelength
  Arms: Low level irradiation

SUMMARY:
The aim of this trial is to show that the low irradiance level is not worse than the high irradiance level in the phototherapy for neonatal jaundice.

DETAILED DESCRIPTION:
Neonatal jaundice is a commonly disease. Phototherapy is performed to prevent from kernicterus.However, light sources and irradiance level are different among hospitals, and it was controversial whether the improvement of jaundice is related to the irradiance level of phototherapy or not. In addition, long-term side effects are not clear, therefore, excessive irradiation should be avoided. The purpose of this study is to show that the low irradiance level is not worse than the high irradiance level in the phototherapy for neonatal jaundice. This study is multicenter randomized controlled trial conducted by Nagoya University Hospital, Anjo Kosei Hospital, Kasugai Municipal Hospital, Handa Hospital, TOYOTA Memorial Hospital, National Hospital Organization Nagoya Medical Center, Japan Red Cross Nagoya Daiichi Hospital, Hekinan Municipal Hospital, and Ogaki Municipal Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Asian full-term neonates with jaundice between 48 and 96 hours of age.

Exclusion Criteria:

* Patients with low-birth-weight, early onset jaundice before 48 hours of age, perinatal asphyxia, antimicrobial therapy or respiratory disorders. Patients with jaundice caused by hemolysis, or functional or anatomic obstruction. Patients who need treatments except for phototherapy.

Ages: 2 Days to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Retreatment rate of neonatal jaundice | one month
  Treatment of neonatal jaundice again after finishing phototherapy.

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Anjo Kosei Hospital, Anjo, Aichi-ken
  - Handa City Hospital, Handa, Aichi-ken
  - Hekinan Municipal Hospital, Hekinan, Aichi-ken
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Japan Red Cross Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - TOYOTA Memorial Hospital, Toyota, Aichi-ken
  - Ogaki Municipal Hospital, Ōgaki, Gifu

IPD SHARING:
Plan to Share IPD: No